CLINICAL TRIAL: NCT04663464
Title: An Open-Label, Randomized, 2-Cohort, 2-Period Crossover Pharmacokinetic Study of Abaloparatide-SC and Abaloparatide-sMTS in Healthy Men and Women
Brief Title: Study to Evaluate and Compare the PK Profiles of Abaloparatide-SC and Abaloparatide-sMTS in a Cohort of Healthy Men and Healthy Women.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Radius Health, Inc. (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BA058-05-024
Record Dates: First submitted 2020-12-04; First posted 2020-12-11 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2020-12

CONDITIONS: Healthy Volunteers
Keywords: osteoporosis; transdermal delivery; solid microstructured transdermal system; abaloparatide; TYMLOS®; abaloparatide-SC; abaloparatide-sMTS; PK
MeSH Terms: conditions — Osteoporosis | interventions — abaloparatide

STUDY DESIGN:
Intervention Model Description: In each of 2 study periods, subjects received receive either a transdermal patch containing 300 μg abaloparatide for 5 minutes or an injection of abaloparatide SC 80 μg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- abaloparatide-SC (Period 1) followed by abaloparatide-sMTS (Period 2) (Experimental): Abaloparatide-SC injection (Period 1) followed by abaloparatide-sMTS application (Period 2). Abaloparatide-SC is a drug-device combination product consisting of abaloparatide, an active synthetic peptide analog of parathyroid hormone related peptide (PTHrP), administered to the periumbilical region via an injection pen. Abaloparatide-sMTS is a drug-device combination product consisting of abaloparatide coated onto a microstructure array for transdermal administration of abaloparatide.
  Interventions: Combination Product: abaloparatide-sMTS; Combination Product: abaloparatide-SC
- Abaloparatide-sMTS (Period 1) followed by abaloparatide-SC (Period 2) (Experimental): Abaloparatide-sMTS (Period 1) application followed by Abaloparatide-SC injection (Period 2).
  Interventions: Combination Product: abaloparatide-sMTS; Combination Product: abaloparatide-SC

INTERVENTIONS:
Combination Product: abaloparatide-sMTS — Single-dose administration of abaloparatide 300 μg applied to the thigh for 5 minutes
  Other Names: BA058; abaloparatide-sMTS
Combination Product: abaloparatide-SC — Single-dose administration of abaloparatide 80 μg subcutaneous injection to the periumbilical region of the abdomen
  Other Names: BA058; abaloparatide-SC

SUMMARY:
A study to evaluate and compare the PK profiles of abaloparatide-SC 80 μg and abaloparatide-sMTS 300 μg in a cohort of healthy men and to make a similar evaluation in a cohort of healthy women

DETAILED DESCRIPTION:
This study aims to evaluate and compare the pharmacokinetic (PK) profiles of abaloparatide-SC 80 μg injected subcutaneously into the periumbilical region of the abdomen, and abaloparatide-sMTS 300 μg applied to the thigh for 5 minutes in a cohort of healthy men and to make a similar evaluation in a cohort of healthy women.

ELIGIBILITY:
Inclusion Criteria

* Male and female subjects aged 40 to 65 years old, inclusive, at Screening;
* Good general health as determined by medical history and physical exam (including vital signs, and has a body mass index between 18 and 32 kg/m^2;
* Laboratory test results within the normal range
* Serum 25-hydroxyvitamin D values must be > 20 ng/mL.

Exclusion Criteria:

* Presence or history of any disorder that may prevent the successful completion of the study;
* Diagnosed with osteoporosis, Paget's disease, or other metabolic bone diseases (eg, vitamin D deficiency or osteomalacia), or had a non-traumatic fracture within 1 year prior to the initial screening;
* History of any cancer within the past 5 years other than squamous or basal cell carcinoma;
* History of allergy to abaloparatide or drugs in a similar pharmacological class;.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-03-27 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
PK Cmax | Time frame for collection of PK data after each single-dose administration, separated by 48 hours
  Maximum observed concentration (Cmax)
PK AUC1 | Time frame for collection of PK data after each single-dose administration, separated by 48 hours
  Area under the plasma concentration-time curve (AUC) from time 0 to the time of the last quantifiable concentration (AUC 0-t)
PK AUC2 | Time frame for collection of PK data after each single-dose administration, separated by 48 hours
  AUC from time 0 extrapolated to time infinity (AUC 0-∞)

SECONDARY OUTCOMES:
Subjects with AEs and SAEs | 10 Days
  Subjects with treatment-emergent AEs and SAEs.

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology, Cincinnati, Ohio, United States